CLINICAL TRIAL: NCT06166511
Title: Evaluation of Laparoscopic Non Anatomical Liver Resection in Hepatic Pathology
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Nader Nasih Adly, Resedent doctor, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Laparoscopic liver resection
Record Dates: First submitted 2023-10-30; First posted 2023-12-12 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Laparoscopic Liver Resection

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group undergo laparoscopic liver resection (Experimental): Any patient from 18 to 65 and has localized liver pathology and underwent laparoscopic non anatomical resection of this pathology
  Interventions: Procedure: Laparoscopic liver resection

INTERVENTIONS:
Procedure: Laparoscopic liver resection — Using Laparoscopy in liver resection

SUMMARY:
Laparoscopy is a type of surgical procedure that allows a surgeon to access the inside of the abdomen and pelvis without making large incisions in the skin.The use of laparoscopy in abdomenal surgeries increases for its great benefits over open surgery as:

1)faster recovery, 2)decrease blood loss, 3)shorter hospital stays, 4)decreased postoperative pain, 5)earlier return to work and resumption of normal daily activity as well as, 6)cosmetic benefits.

few studies discuss the efficacy and safety of using Laparoscopy in liver non anatomical resection.

DETAILED DESCRIPTION:
this study will include any male and female above 18 that presented with localized liver pathology (as benign hepatic tumours, resectable primary(HCC) or secondary malignancies, hydatid cyst any other hepatic cysts, haemangiomas,etc…...) and underwent laparoscopic non anatomical resection of liver in Assiut university hospitals. Investigators will record the time of operation, number of cases with intra operative mortality or complication and then follow up these patients during time of hospital stay for:

1) post operative pain 2) secondary bleeding and 3) wound infection.

Then follow up these patients in out patient clinic visit for their:

1. satisfaction
2. cosmetic outcomes and
3. rate of recurrence of the pathology.

ELIGIBILITY:
Inclusion Criteria:

* any male or female above 18 that has one of the following pathologies and underwent non anatomical hepatic resection:
* hepatic benign tumours as adenoma
* resectable secondary malignancies (2)
* any type of hepatic cysts e.g., hydatid cyst
* HCC on top of liver cirrhosis.

Exclusion Criteria:

* 1) any immunocompromised patient 2) Patient with contraindicdtions to use laparoscopy. 3) patient who are difficult to follow up.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-01-10 (Estimated); Primary Completion 2025-03-10 (Estimated); Study Completion 2025-05-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of intra operative mortality | 2 years
  Number of cases die intra operative
Length of operation | 2 years
  Time of operation
Post operative pain | 2 years
  Pain scale post operative
Incidence of intra operative complications | 2 years
  Type of complications and Its incidence
Length of hospital stay | 2 years
  Time spended by cases in hospital
Incidence of post operative complications | 2 years
  Type and incidence of post operative complications

SECONDARY OUTCOMES:
Cosmetic outcome | 2 years
  Patient cosmetic sutisfacton
Incidence of recurrence of pathology | 2 years
  Number of cases with same pathology recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Nader N Adly, Principal Investigator — Assuit University hospitals
Locations (1):
- Assuit University hospitals, Asyut, Assuit, Egypt

REFERENCES:
- [Background] Garlipp B, Gibbs P, Van Hazel GA, Jeyarajah R, Martin RCG, Bruns CJ, Lang H, Manas DM, Ettorre GM, Pardo F, Donckier V, Benckert C, van Gulik TM, Goere D, Schoen M, Pratschke J, Bechstein WO, de la Cuesta AM, Adeyemi S, Ricke J, Seidensticker M. Secondary technical resectability of colorectal cancer liver metastases after chemotherapy with or without selective internal radiotherapy in the randomized SIRFLOX trial. Br J Surg. 2019 Dec;106(13):1837-1846. doi: 10.1002/bjs.11283. Epub 2019 Aug 19. PMID 31424576